CLINICAL TRIAL: NCT02083627
Title: A Phase 1, Open Label, Randomized, Two-way Crossover Study to Evaluate the Effect of Multiple Doses of Fidaxomicin on the Single Dose Pharmacokinetics of Rosuvastatin in Healthy Male Subjects
Brief Title: A Study to Assess the Effects of Multiple Doses of Fidaxomicin on a Single Dose of Rosuvastatin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2819-CL-2003; 2012-003924-20 (EudraCT Number)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Drug-Drug Interaction (DDI); Intestinal Absorption; Healthy Subjects; Pharmacokinetics of Rosuvastatin; Pharmacokinetics of Fidaxomicin
Keywords: Pharmacokinetics; Drug-Drug Interaction; Intestinal Absorption; Fidaxomicin; Rosuvastatin; Multiple Doses; Single Doses
MeSH Terms: interventions — Rosuvastatin Calcium; Fidaxomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:Single rosuvastatin,multiple fidaxomicin,single rosuvastatin (Experimental)
  Interventions: Drug: rosuvastatin; Drug: fidaxomicin
- 2:Multiple fidaxomicin,single rosuvastatin,single rosuvastatin (Experimental)
  Interventions: Drug: rosuvastatin; Drug: fidaxomicin

INTERVENTIONS:
Drug: rosuvastatin — Oral
  Other Names: Crestor®
Drug: fidaxomicin — Oral
  Other Names: Dificlir™; DIFICID®

SUMMARY:
This study will assess the effect of multiple doses of fidaxomicin on the single dose pharmacokinetics of rosuvastatin in healthy male subjects. Determine the safety and tolerability of multiple doses of fidaxomicin in the presence of a single dose of rosuvastatin in healthy male subjects. Also determine the pharmacokinetics of multiple doses of fidaxomicin and its metabolite OP-1118.

DETAILED DESCRIPTION:
Sequence 1:

Thirteen subjects receive an oral dose of rosuvastatin on Day 1 in Period 1 and on Day 13 in Period 2 and twice-daily oral doses of fidaxomicin on Days 8 to 17 in Period 2, according to the following treatment schedule:

* Period 1: Subjects receive a single oral dose of rosuvastatin on Day 1, followed by a 5-day pharmacokinetic (PK) sampling period.
* Period 2: The same subjects receive fidaxomicin twice daily for 5 days (Days 8 to 12). On Day 13, a single oral dose of rosuvastatin and an oral dose of fidaxomicin is administered simultaneously in the morning. Twice-daily treatment with fidaxomicin continues until the end of Day 17. Subjects are discharged on Day 18 when all assessments are performed and if there are no medical reasons to prolong the stay.

Sequence 2:

Thirteen subjects receive an oral dose of rosuvastatin on Day 6 in Period 1 and on Day 14 in Period 2. Oral doses of fidaxomicin are administered twice daily for 10 days in Period 1, according to the following treatment schedule:

* Period 1: Subjects receive fidaxomicin twice daily for 5 days (Days 1 to 5). On Day 6, a single oral dose of rosuvastatin is administered simultaneously with an oral dose of fidaxomicin in the morning. Twice daily treatment with fidaxomicin continues until the end of Day 10.
* Period 2: Subjects receive a single oral dose of rosuvastatin on Day 14, followed by a 5-day PK sampling period. Subjects are discharged on Day 19 when all assessments are performed and if there are no medical reasons to prolong the stay.

In both sequences, subjects return to the clinical unit for an End of Study Visit (ESV) 7 to 14 days after (early) discharge.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a Body Mass Index (BMI) range of 18.5 to 30.0 kg/m2. The subject weighs at least 50 kg at Screening.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 90 days after final study drug administration.
* The subject must not donate sperm starting at Screening and through-out the study period and for at least 90 days after final study drug administration.

Exclusion Criteria:

* The subject has a history of or current Clostridium difficile infection.
* The subject has a history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
* The subject has an irregular defecation pattern.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Effect of multiple doses of fidaxomicin on the single dose pharmacokinetics of rosuvastatin as measured by maximum observed concentration | Day 1-6 (sequence1/period1) & Day 13-18 (sequence1/period2) Day 6-11 (sequence2/period1) & Day 14-19 (sequence2/period2)
  Cmax (maximum observed concentration)
Effect of multiple doses of fidaxomicin on the single dose pharmacokinetics of rosuvastatin as measured by area under the concentration time curve from time zero extrapolated to infinity | Day 1-6 (sequence1/period1) & Day 13-18 (sequence1/period2) Day 6-11 (sequence2/period1) & Day 14-19 (sequence2/period2)
  AUCinf (area under the concentration time curve from time zero extrapolated to infinity)

SECONDARY OUTCOMES:
Effect of multiple doses of fidaxomicin on the single dose pharmacokinetic profile of rosuvastatin | Day 1-6 (sequence1/period1) & Day 13-18 (sequence1/period2) Day 6-11 (sequence2/period1) & Day 14-19 (sequence2/period2)
  AUClast (Area under the concentration time curve from time point zero to last quantifiable concentration), CL/F (apparent clearance following oral administration), tmax (time to attain Cmax (maximum observed concentration), t1/2 (terminal elimination half-life), Vz/F (apparent volume of distribution during terminal phase)
Safety and tolerability of multiple doses of fidaxomicin in the presence of a single dose of rosuvastatin | Screening (Day -22 to -2) to ESV (7 to 14 days after (early) discharge)
  Adverse Events (AE), vital signs, laboratory tests, 12-lead Electrocardiogram (ECG)
PK of multiple doses of fidaxomicin and its metabolite OP-1118 | Day 9-15 (sequence 1/period2) & Day 2-8 (sequence2/period1)
  tmax (time to attain Cmax (maximum observed concentration), AUCtau (area under the concentration time curve over a dosing interval), Ctrough (measured concentration at the end of a dosing interval (taken directly before next administration))

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel GmbH, Berlin, Germany